CLINICAL TRIAL: NCT07030972
Title: Investigation of the Effect of Deep Friction Massage Applied to Patients With Bicipital Tendinitis on Pain, Functional Capacity, Kinesiophobia, and Quality of Life
Brief Title: Effect of Deep Friction Massage on Pain, Function, Kinesiophobia, and Quality of Life in Bicipital Tendinitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Muharrem Gökhan Beydağı, Assistant Professor, PT, PhD, Firat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FU_MGBeydagi_Omuz_B_2025/06-39
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Bicipital Tendonitis
Keywords: bicipital tendinitis; deep friction massage
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The type of the research is a parallel randomized controlled trial with before-after measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Individuals in the control groups will be included in a routine exercise program. This exercise program will include shoulder joint range of motion exercises, finger ladder, Codman, and stick exercises, which will be applied to maintain functional range of motion in the early stages and increase it in the later stages. Isometric exercises will be applied to the scapular muscles to maintain muscle strength in the early stages. In the later stages, rotator cuff, scapular stabilizer, and deltoid strengthening exercises will be demonstrated and applied. Low-resistance therabands will be used for strengthening at the beginning. Additionally, neuromuscular control exercises and proprioceptive exercises will be included in the treatment to enhance joint stabilization and coordination. The exercises will be performed over a 6-week period, 3 days per week, with 10-30 repetitions.
  Interventions: Other: Exercise
- Intervention group (Experimental): Individuals in the intervention group will receive deep friction massage on the biceps tendon in addition to the routine exercise program and following the exercise program. The individual will be placed in a long sitting position with their back supported. While the patient's shoulder is next to the body and the elbow is flexed at 90 degrees, the therapist's thumb will be placed on the painful area on the extension of the biceps tendon fibers and a deep friction massage will be applied to the point where the tendonitis occurs in a transverse direction for 3-10 minutes.
  Interventions: Other: Exercise; Other: Deep friction massage

INTERVENTIONS:
Other: Exercise — Individuals in the control and intervention groups will be included in a routine exercise program. For this exercise program; shoulder joint range of motion exercises, finger ladder, Codman and stick exercises will be given to protect functional range of motion in the early stages and to increase it in the later stages. Isometric exercises will be performed on the scapular muscles in the early stages to preserve muscle strength. In the later stages, rotator cuff, scapula stabilizers and deltoid strengthening exercises will be shown and applied, initially with low-resistance therabants for strengthening. In addition, neuromuscular control exercises and proprioceptive exercises will be included in the treatment to increase joint stabilization and coordination. Exercises will be performed for 6 weeks, 3 days a week, with 10-30 repetitions.
Other: Deep friction massage — Individuals in the intervention group will receive a deep friction massage to the biceps tendon after the exercise program. The individual will be placed in a long sitting position with their back supported. While the patient's shoulder is next to the body and the elbow is flexed at 90 degrees, the therapist's thumb will be placed on the painful area on the extension of the biceps tendon fibers and a deep friction massage will be applied to the point where the tendonitis occurs in a transverse direction for 3-10 minutes.
  Arms: Intervention group

SUMMARY:
Bicipital tendinitis is a condition caused by inflammation of the biceps tendon, resulting in pain and limited movement in the front of the shoulder. This condition usually develops due to repetitive shoulder movements or overuse and can negatively affect daily life.

Treatment usually involves medications, cold applications, rest, and exercises. However, in some cases, these methods may not be sufficient. This study aims to investigate the effects of deep friction massage (DFM) when applied in addition to a standard exercise program. DFM is a massage technique that supports tissue healing, reduces pain, and improves mobility.

Within the scope of the study, the effects of DFM combined with exercise on pain, functional capacity, fear of movement (kinesiophobia), and quality of life will be evaluated. The findings obtained aim to contribute to the development of more effective approaches in the treatment of biceps tendinitis.

DETAILED DESCRIPTION:
Bicipital tendinitis is a condition characterized by inflammation of the long head of the biceps tendon, causing pain and tenderness in the front of the shoulder. It typically develops due to repetitive shoulder movements or overuse and, if left untreated, can negatively impact quality of life. Treatment for biceps tendinitis focuses on reducing inflammation and swelling, strengthening the tendon, and preventing tendon rupture. Early/initial treatments for biceps tendinitis include nonsteroidal anti-inflammatory drugs, activity modification, nonsteroidal anti-inflammatory gels or patches for pain, and cold applications for pain and swelling. If symptoms do not improve, physical therapy may be recommended. These treatments typically include stretching and strengthening exercises, massage, or ultrasound therapy. Exercises aim to help keep muscles, joints, and tendons mobile and flexible. If symptoms are severe or persistent despite initial/early treatment, the doctor may recommend a steroid injection into the affected area to reduce inflammation and pain. After the injection, patients are typically prescribed rest, ice, acetaminophen (Tylenol) for pain, and a regimen of stretching/strengthening exercises.

Another important treatment method in the conservative management of tendinopathies is Deep Friction Massage (DFM). DFM is an approach that mechanically supports the remodeling of tissue and the healing process. This technique helps meet the tendon's oxygen and nutrient requirements by increasing blood flow in the treated area, while supporting the alignment of collagen fibers and facilitating the reorganization of scar tissue. The effects of deep friction massage on pain reduction and functional capacity improvement have been extensively documented in the literature. Additionally, the positive effects of this method on flexibility and range of motion from a biomechanical perspective are one of the reasons it is preferred in the management of musculoskeletal disorders.

The investigators believe that the application of deep friction massage in addition to a standard exercise program in patients with bicipital tendinitis could be a useful combination therapy to support tendon healing. This approach may create a synergistic effect in tendon healing by combining the positive effects of exercise with the long-term tissue benefits of deep friction massage. There are a limited number of studies in the literature suggesting that this combination is effective; therefore, more comprehensive and controlled research is needed to guide clinical practice.

Pain, functional capacity, kinesiophobia (fear of movement), and quality of life are critical in assessing the effects of biceps tendinitis on patients. Improving these parameters can accelerate patients' return to daily activities and improve their overall health. In light of this information, it is thought that the combined application of an exercise program and deep friction massage could be considered a potential treatment strategy for pain management and functional improvement in the treatment of biceps tendinitis. This study aims to evaluate the effects of deep friction massage, applied in addition to an exercise program, on pain, functional capacity, kinesiophobia, and quality of life in patients with biceps tendinitis. This will provide further insight into the efficacy of combined treatment methods and guide clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bicipital tendinitis (tendinosis)
* Be between 20 and 55 years of age
* Have shoulder pain lasting longer than 3 months

Exclusion Criteria:

* Shoulder impingement or frozen shoulder
* Another shoulder problem such as a full-thickness rotator cuff tear or instability
* Having received physical therapy or manual therapy for the same shoulder within the past year
* History of upper extremity fracture
* History of shoulder surgery
* Presence of entrapment neuropathy
* Having radicular pain originating from the cervical vertebrae
* Having a systemic musculoskeletal disease
* Having mental and cognitive problems

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | before-after treatment (baseline, 6th week and 12th week)
  The Visual Analog Scale (VAS) will be used to determine the intensity of pain and to compare the pain felt before and after treatment (baseline, 6th week and 12th week). VAS is a reliable and easily applicable test used to measure values that cannot be easily measured numerically by converting them into a numerical format. The lowest and highest definitions of the parameters to be evaluated are written on both ends of a 100 mm line. The patient is asked to mark the most appropriate value (location) between these two extreme points. When this scale is used for pain, the numbers "0" are written on one end to indicate no pain and "10" are written on the other end to indicate the most severe pain, and this is converted into a template, numbers between 0-10 are placed on the line and the patient is asked to choose the closest number.

SECONDARY OUTCOMES:
Assessment of Functional Capacity | before and after treatment (at baseline, 6 weeks, and 12 weeks)
  Individuals' functional capacities will be assessed using the Shoulder, Arm, and Hand Problems Short Form (Q-DASH).
  Shoulder, Arm, and Hand Problems Short Form (Q-DASH):
  The Quick DASH questionnaire, which is the short form of the Shoulder, Arm, and Hand Problems (DASH-T) questionnaire validated and tested for reliability in Turkish by Düger et al. (2006), will be used. The 11-item questionnaire subjectively assesses the functional status of the upper extremity using a Likert scale. Patients will be asked to complete the questionnaire themselves, and the total score obtained will be converted into a total score ranging from 0 to 100 using a formula developed for the questionnaire (Gummesson et al. 2004). Values closer to 0 indicate good functional outcomes.

OTHER OUTCOMES:
Assessment of Normal Joint Movement | pre- and post-treatment (baseline, 6 weeks, and 12 weeks)
  Individuals' normal shoulder joint range of motion will be measured using a digital goniometer. The active and passive range of motion of the shoulder in extension, flexion, abduction, adduction, internal, and external rotation will be assessed. The normal range of motion of the affected shoulder will be evaluated. Each test will be performed three times to ensure accuracy, and the average of the three measurements will be recorded.
Evaluation of Kinesiophobia | before and after treatment (at baseline, week 6, and week 12)
  The short form of the Tampa Kinesiophobia Scale (TKÖ) will be used to assess individuals' kinesiophobia levels. The TKÖ is a measure developed in 1991 by Miller, Kopri, and Todd, but later republished by Vlaeyen et al., and used to assess fear of movement. The TKÖ consists of 17 questions. It includes questions related to injury/re-injury and fear-avoidance situations in work-related activities, and individuals answer them themselves. It is scored on a four-point Likert scale (1 = strongly disagree, 4 = strongly agree). At the end of the scale, a score between 17 and 68 is obtained, and high scores are defined as kinesiophobia.
Assessment of Quality of Life | before and after treatment (at baseline, week 6, and week 12)
  The SF-12 questionnaire will be used to assess individuals' quality of life. Ware et al. (1995) developed a shortened version of the SF-36 quality of life questionnaire. Soylu et al. (2022) also examined the validity and reliability of the SF-12 Quality of Life Scale in Turkish. The SF-12 is a questionnaire used to assess individuals' general health status, physical and psychological functions, social activities, and quality of life. It consists of 12 questions, and the general health score is calculated based on the answers given to these questions. Thanks to the SF-12, the 36 items were reduced to 12 items, allowing participants to complete the questionnaire in less than one-third of the time spent on the SF-36. Ware demonstrated a strong correlation between the two tools, showing that approximately 90% of the variability in both the physical and mental component summaries of the SF-36 is explained by the same summary mea

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat Üniversitesi, Elâzığ, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size and ethical restrictions regarding patient confidentiality in this single-center study, individual participant data will not be publicly shared. However, aggregated data will be available upon reasonable request.

REFERENCES:
- [Result] Bozgeyik S, Kinikli GI, Topal Y, Beydagi MG, Turhan E, Kilinc HE, Guney-Deniz H. Supervised exercises have superior effects compared to home-based exercises for patients with knee osteoarthritis following platelet-rich plasma injection. Res Sports Med. 2024 Mar-Apr;32(2):279-289. doi: 10.1080/15438627.2022.2102920. Epub 2022 Jul 19. PMID 35854659